CLINICAL TRIAL: NCT03885102
Title: Exercise During Hemodialysis: The Dialysis Training Therapy (DiaTT) Trial
Brief Title: Dialysis Training Therapy: The DiaTT Trial
Acronym: DiaTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. med. Martin Halle (Other)
Collaborators: Technical University of Munich (Other); University Hospital of Cologne (Other); KfH Kuratorium für Dialyse und Nierentransplantation (Unknown); Clinical Trials Unit Freiburg (Other); AOK PLUS (Industry); BARMER (Other); Techniker Krankenkasse (Other); Federal Joint Committee (Other Government)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Martin Halle, Univ.-Prof. MD, Technical University of Munich
Organization: Technical University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 509/18S-KK
Record Dates: First submitted 2019-03-18; First posted 2019-03-21 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Chronic Kidney Diseases; Hemodialysis
Keywords: chronic kidney disease; hemodialysis; intradialytic exercise; physical activity; safety; health economics; health literacy; training therapy
MeSH Terms: conditions — Renal Insufficiency, Chronic; Motor Activity

STUDY DESIGN:
Intervention Model Description: Random assignment in 1:1 ratio into either intervention group (12 months intradialytic exercise intervention; 50% aerobic exercise, 50% resistance training; thrice a week for 60 min per dialysis session) and health literacy counselling (HLC) or control group/usual care (Usual care without any exercise intervention or HLC)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 12 months intradialytic exercise intervention
  Interventions: Behavioral: Intradialytic exercise intervention
- Usual care (Active Comparator): Usual care according to current guidelines
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Intradialytic exercise intervention — 50% aerobic exercise, 50% resistance training thrice a week for 60 min per dialysis session, and health literacy counselling
  Arms: Intervention
Behavioral: Usual Care — Usual care with no exercise intervention or health literacy counselling
  Arms: Usual care

SUMMARY:
DiaTT is an interventional, cluster-randomized (1:1), multicenter trial for patients with chronic kidney disease undergoing hemodialysis (n=1,100). This trial will test the effectiveness (by change of sit-to-stand test between baseline and 12 months) of intradialytic exercise training (ET) and health literacy counseling (HLC) for 12 months (Intervention group) in comparison to control group (usual care, UC; no ET, no HLC).

DETAILED DESCRIPTION:
The primary objective of this trial is to assess the effectiveness of intradialytic exercise training (ET) and health literacy counselling (HLC) over 12 months intervention in patients undergoing chronic outpatient hemodialysis as compared to usual care (UC). The primary endpoint is change in Sit-to-Stand (STS60) test, from baseline to after 12 months intervention. The ET consists of both resistance and endurance training, focusing on improving patients' health status and physical functioning. Health literacy counseling aims at improving education, proficiency and self-awareness of the patient.

All patients undergoing hemodialysis in participating centers (clusters) for at least four weeks are eligible to participate in the study. Irrespective of randomized center (cluster) group assignment, all dialysis and overall medical treatments will remain unchanged and follow standard of care and center routine without adaptations to the training intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age
* chronic ambulatory hemodialysis for > 4 weeks
* Written and signed confirmation by the treating dialysis physician that the patient is able to exercise
* signed informed consent to participation in QiN registry
* signed informed consent obtained according to confidentiality and data protection regulation, international guidelines and local laws

Exclusion Criteria:

* Unstable angina pectoris
* Uncontrolled arterial hypertension (systolic blood pressure > 180 mmHg or diastolic BP > 105 mmHg on repeated measurements)
* Uncontrolled tachycardia
* Acute severe infection
* Planned live kidney transplantation within the next 12 months
* Planned conversion to home-hemodialysis or peritoneal dialysis within the next 12 months
* Dialyzing in long overnight dialysis shift
* Participation in a regular exercise program during hemodialysis sessions (≥ 1/week) in the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1211 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Sit-to-stand test (STS60) | between baseline and 12 months
  Change of Sit-to-stand test (STS 60) (number of repetitions in 60 seconds)

SECONDARY OUTCOMES:
Overall survival | 12 months
  Defined as time from center randomization until death from any cause, or as time from center randomization until the patient was last alive (censored observations).
3-point MACE | 12 months
  a composite of cardiovascular death, non-fatal stroke, or non-fatal myocardial infarction
sudden death | 12 months
  Patients alive will be considered as censored observations, and death from other causes will be considered as a competing event
Sit-to-stand test (STS60) | 3, 6 and 9 months
  measured in number of repetitions in 60 seconds
Timed-up-and-go test (TUG) | 3, 6, 9, and 12 months
  measured in time (seconds)
Six-Minutes-Walk test (6MWT) | 3, 6, 9, and 12 months
  measured in distance (meter)
Grip strength test (GST) | 3, 6, 9, and 12 months
  measured in kilogram
hospitalizations | 12 months
  measured in number and days of hospitalization for comorbidities
frailty by Multidimensional Prognostic Index (MPI) | 3,6 and 12 months
  measured in change of scale in questionnaire
Serum phosphate | 3, 6, 9 and 12 months
  measured in mmol/L
Erythropoietin dose | 3, 6, 9, and 12 months
  measured in IE/week
Quality of life by SF-36 | 3, 6 and 12 months
  measured in change of scale by questionnaire
Health literacy by HLS-EU-Q16 | 3, 6 and 12 months
  measured in change of scale in questionnaire
health economics by medication | 12 months
  measured in total costs between between study arms
health economics by hospitalization | 12 months
  measured in days in hospital between between study arms
health economics by transportation | 12 months
  measured in total costs between between study arms
health economics by medical assistance tools | 12 months
  measured in total costs between between study arms
health economics by nursing | 12 months
  measured in total costs between between study arms
health economics by sick leave from workplace | 12 months
  measured in days between between study arms
needle dislocation/ catheter disconnection | 12 months
  number of dialysis needle dislocation/ dialysis catheter disconnection
symptomatic hypotensive episodes | 12 months
  number of symptomatic hypotensive episodes
cramps | 12 months
  number of cramps

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Ihorst, PhD, Study Chair — Clinical Trials Unit Freiburg, Medical Center, University of Freiburg; Gero von Gersdorff, MD, Study Chair — Department II of Internal Medicine, University of Cologne; Kirsten Anding-Rost, MD, Study Chair — KfH Kuratorium für Dialyse und Nierentransplantation e.V.; Martin Halle, Prof. MD, Principal Investigator — Department of Prevention, Rehabilitation and Sports medicine, University hospital 'Klinikum rechts der Isar', Technical University of Munich
Locations (21):
- Germany (21):
  - KfH-Nierenzentrum, Amberg, Bavaria
  - KfH-Nierenzentrum, Aschaffenburg, Bavaria
  - KfH-Nierenzentrum, Bamberg, Bavaria
  - KfH-Nierenzentrum, Coburg, Bavaria
  - KfH-Nierenzentrum, Dachau, Bavaria
  - KfH-Nierenzentrum, Ebersberg, Bavaria
  - KfH-Nierenzentrum, Freising, Bavaria
  - KfH-Nierenzentrum, Fürstenzell, Bavaria
  - KfH-Nierenzentrum, Fürth, Bavaria
  - KfH-Nierenzentrum, München, Bavaria
  - KfH-Nierenzentrum, Straubing, Bavaria
  - KfH-Nierenzentrum, Aachen, Northrhine
  - KfH-Nierenzentrum, Bergisch Gladbach, Northrhine
  - KfH-Nierenzentrum, Cologne, Northrhine
  - KfH-Nierenzentrum, Halle, Saxony-Anhalt
  - KfH-Nierenzentrum, Magdeburg, Saxony-Anhalt
  - KfH-Nierenzentrum, Jena, Thuringia
  - KfH-Nierenzentrum, Sonneberg, Thuringia
  - KfH-Nierenzentrum, Bochum, Westphalia
  - KfH-Nierenzentrum, Hagen, Westphalia
  - KfH-Nierenzentrum, Marl, Westphalia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] von Gersdorff G, von Korn P, Duvinage A, Ihorst G, Josef A, Kaufmann M, Baer T, Fellerhoff T, Fuhrmann I, Koesel E, Zeissler S, Bobka L, Heinrich M, Schindler A, Weber R, Breuer C, Meyer AM, Polidori MC, Dinges SMT, Schoenfeld J, Siebenbuerger M, Degenhardt S, Anding-Rost K, Halle M. Cluster Randomized Controlled Trial on the Effects of 12 Months of Combined Exercise Training during Hemodialysis in Patients with Chronic Kidney Disease-Study Protocol of the Dialysis Training Therapy (DiaTT) Trial. Methods Protoc. 2021 Aug 31;4(3):60. doi: 10.3390/mps4030060. PMID 34564306
- [Derived] Anding-Rost K, von Gersdorff G, von Korn P, Ihorst G, Josef A, Kaufmann M, Huber M, Bar T, Zeissler S, Hofling S, Breuer C, Gartner N, Haykowsky MJ, Degenhardt S, Wanner C, Halle M. Exercise during Hemodialysis in Patients with Chronic Kidney Failure. NEJM Evid. 2023 Sep;2(9):EVIDoa2300057. doi: 10.1056/EVIDoa2300057. Epub 2023 Jun 17. PMID 38320198